CLINICAL TRIAL: NCT00774761
Title: A Randomized, Multiple-Dose,Double-Blind,Crossover Trial to Assess the Systemic Exposure of Fluticasone Propionate (FP)/Formoterol Fumarate (FF) Fixed-Dose Combination in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study Evaluating Systemic Exposure and Pharmacodynamics in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 191-087
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic; Obstructive; Pulmonary; Disease; COPD; Pharmacodynamic; Pharmacokinetic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Disease | interventions — Fluticasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: fluticasone propionate/formoterol fumarate
- 2 (Experimental)
  Interventions: Drug: fluticasone propionate/formoterol fumarate
- 3 (Active Comparator)
  Interventions: Drug: fluticasone propionate
- 4 (Active Comparator)
  Interventions: Drug: fluticasone propionate
- 5 (Active Comparator)
  Interventions: Drug: formoterol fumarate

INTERVENTIONS:
Drug: fluticasone propionate/formoterol fumarate — inhalation suspension
  Arms: 1; 2
Drug: fluticasone propionate — inhalation suspension
  Arms: 3; 4
Drug: formoterol fumarate — inhalation solution
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the systemic exposure and pharmacodynamics of two doses of nebulized fluticasone/formoterol combination as compared to the monocomponents.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the requirements of the study and provide consent
* Medical diagnosis of COPD
* A current or prior history of at least 10-pack years of cigarette smoking
* Female of child-bearing potential to use adequate birth control

Exclusion Criteria:

* Diagnosis of asthma
* Other significant disease than COPD
* Has donated a unit of blood within 30 days of study, or intends to donate
* QTc greater than 0.460 seconds
* Subjects who had radiation or chemotherapy in the previous 12 months
* Subjects who had lung resection
* History of illegal drug abuse or alcohol abuse within the past 5 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Plasma AUC(0-t) after 1 week of dosing | PK sampling over 24 hrs

SECONDARY OUTCOMES:
FEV1 | pre-dose and 2 hrs post-dose

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Investigative Site, San Diego, California
  - Investigative Site, Panama City, Florida
  - Investigative Site, Madisonville, Kentucky
  - Investigative Site, Sunset, Louisiana
  - Investigative Site, Charlotte, North Carolina
  - Investigative Site, Medford, Oregon
  - Investigative Site, Greenville, South Carolina
  - Investigative Site, Spartanburg, South Carolina
  - Investigative Site, Union, South Carolina
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Spokane, Washington
  - Investigative Site, Tacoma, Washington